CLINICAL TRIAL: NCT00650780
Title: Vitamin D Binding Protein (Gc) Allele Variation Effects Response to Vitamin D Treatment
Acronym: Gc
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Laura Armas, Creighton University
Other Study IDs: Creighton4
Record Dates: First submitted 2008-03-30; First posted 2008-04-02 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Vitamin D Status
Keywords: Viatmin D, 25-hydroxyvitamin D, Vitamin D binding protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All of the subjects will have measurements of Gc concentration and phenotype

SUMMARY:
We have just completed a randomized, clinical trial of 100,000 IU Vitamin D3 given as a single dose at the beginning of winter. We found a wide range of responses to the dose. This study proposes that genetic differences account for some of the variation in response of 25(OH)D levels after treatment with oral Vitamin D.

DETAILED DESCRIPTION:
We suspect that the wide range of response is effected by other factors such as variation in Vitamin D binding protein (the major transporter of Vitamin D metabolites).

Gc, also known as Vitamin D binding protein (DBP), group specific component, or Gc globulin, is a 52-58 kDa multifunctional plasma protein, synthesized in the liver. The gene encoding for Gc is located on chromosome 4, and three common co-dominant alleles give rise to three phenotypes (Gc1s, Gc1f, and Gc2). Gc binds actin, recruits neutrophil leukocytes and converts into a macrophage- and osteoclast- activating factor. It also is the major transporter of Vitamin D and its' metabolites. Lauridsen et al. showed that Gc phenotype correlates with 25(OH)D levels in a group of postmenopausal women.

This study proposes that Gc phenotype accounts for some of the variation in response of 25(OH)D levels after treatment with oral Vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to participate with an additional blood draw.
* Must have been in the previous study.

Exclusion Criteria:

* Will not be eligible if not a part of the previous study

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include thirty males and females who took part in a previous study of a single oral dose of vitamin D.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Gc concentration and phenotype | at 1st visit

CONTACTS AND LOCATIONS:
Overall Officials: Laura Armas, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States